CLINICAL TRIAL: NCT02486042
Title: Omega-3 Long Chain Polyunsaturated Fatty Acid (LCPUFA) Supplementation in Very Low Birth Weight Infants for The Prevention Retinopathy of Prematurity: Proposal for a Prospective Randomized Controlled Masked Clinical Trial With Lipidomic and Transcriptomic Analyses
Brief Title: Omega-3 Long Chain Polyunsaturated Fatty Acid (LCPUFA) Supplementation in Very Low Birth Weight Infants for The Prevention Retinopathy of Prematurity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: The Hartwell Foundation (Other)
Responsible Party: Principal Investigator, Shira Robbins, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 140253
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Results first posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-11

CONDITIONS: Retinopathy of Prematurity
Keywords: ROP; Premature infant
MeSH Terms: conditions — Retinopathy of Prematurity; Premature Birth | interventions — fish oil triglycerides; Docosahexaenoic Acids; soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Standard Nutrition) (Active Comparator): Infants in this group will receive standard lipids (predominantly Omega-6 fatty acids).
  Interventions: Dietary Supplement: Standard lipids (primarily omega-6 fatty acids)
- Omegaven (Experimental): Infants in this group will receive lipid supplementation with omega-3 fatty acids.
  Interventions: Drug: Omegaven

INTERVENTIONS:
Drug: Omegaven — Infants will receive nutritional supplementation with omega-3 fatty acids (omegaven).
  Other Names: Omega-3
  Arms: Omegaven
Dietary Supplement: Standard lipids (primarily omega-6 fatty acids) — Infants will receive nutritional supplementation with standard intralipid, composed primarily of omega-6 fatty acids.
  Other Names: Intralipid
  Arms: Standard of Care (Standard Nutrition)

SUMMARY:
Retinopathy of prematurity (ROP) is a blinding disease affecting infants born prematurely. These infants do not have enough essential fatty acids to structurally support the retina, the nerve tissue in the eye which allows us to see. A recent study showed that giving omega-3 (n-3) fatty acids to these infants soon after birth made them less likely to need invasive treatments for eye disease. This research trial will give young infants born prematurely n-3 fish oil treatment and look at how this changes factors in the blood that promote disease. Detailed blood studies comparing infants with and without ROP will be performed and the infants will be followed over time to assess their eye development.

DETAILED DESCRIPTION:
Approximately 517,000 infants are born prematurely every year. As low birth weight and premature infants are surviving longer, they are at risk of developing severe retinopathy of prematurity (ROP).

ROP is a disease of the eye affecting prematurely-born babies. It is thought to be caused by disorganized growth of retinal blood vessels which may result in scarring and retinal detachment. ROP can be mild and may resolve spontaneously, but it may lead to blindness in serious cases. ROP is the leading cause of irreversible childhood blindness in the United States. As such, all preterm babies are at risk for ROP, and very low birth weight is an important risk factor.

Researchers have found that increasing omega-3 fatty acids and decreasing omega-6 fatty acids in the diet of mice with eye disease similar to ROP had reduced areas of blood vessel loss and abnormal blood vessel growth. These findings represent new evidence suggesting the possibility that omega-3 fatty acids act as protective factors in diseases that affect retinal blood vessels.

Omega-3 fatty acids make compounds that protect against the growth of abnormal blood vessels by preventing inflammation.

In two European studies, this treatment decreased the risk of needing laser treatment in the eye for ROP. This study has not yet been repeated in the United States. The purpose of this study is to learn how omega-3 fatty acid supplementation in low birth weight infants changes the blood profile of infants receiving this nutritional treatment.

Infants are enrolled in this study shortly after birth and receive IV and/or oral supplementation until they are full term or the retinal blood vessels have completely developed, shortly after term. Once the treatment is over, these infants will continue to be followed for growth and development of their eyes.

ELIGIBILITY:
Inclusion Criteria:

* Infants born less than or equal to 30 weeks gestation or less than 1500 g at birth

Exclusion Criteria:

* Patients with liver disease as tested by liver function tests (LFTs)
* ≤ 500 grams birthweight

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2014-03; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shira L. Robbins, M.D., Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego Jacobs Medical Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gould JF, Smithers LG, Makrides M. The effect of maternal omega-3 (n-3) LCPUFA supplementation during pregnancy on early childhood cognitive and visual development: a systematic review and meta-analysis of randomized controlled trials. Am J Clin Nutr. 2013 Mar;97(3):531-44. doi: 10.3945/ajcn.112.045781. Epub 2013 Jan 30. PMID 23364006
- [Background] Clandinin MT, Chappell JE, Heim T, Swyer PR, Chance GW. Fatty acid utilization in perinatal de novo synthesis of tissues. Early Hum Dev. 1981 Sep;5(4):355-66. doi: 10.1016/0378-3782(81)90016-5. PMID 7285840
- [Background] Arsic A, Vucic V, Prekajski N, Tepsic J, Ristic-Medic D, Velickovic V, Glibetic M. Different fatty acid composition of serum phospholipids of small and appropriate for gestational age preterm infants and of milk from their mothers. Hippokratia. 2012 Jul;16(3):230-5. PMID 23935289
- [Background] Pawlik D, Lauterbach R, Walczak M, Hurkala J, Sherman MP. Fish-oil fat emulsion supplementation reduces the risk of retinopathy in very low birth weight infants: a prospective, randomized study. JPEN J Parenter Enteral Nutr. 2014 Aug;38(6):711-6. doi: 10.1177/0148607113499373. Epub 2013 Aug 20. PMID 23963690
- [Background] Connor KM, SanGiovanni JP, Lofqvist C, Aderman CM, Chen J, Higuchi A, Hong S, Pravda EA, Majchrzak S, Carper D, Hellstrom A, Kang JX, Chew EY, Salem N Jr, Serhan CN, Smith LEH. Increased dietary intake of omega-3-polyunsaturated fatty acids reduces pathological retinal angiogenesis. Nat Med. 2007 Jul;13(7):868-873. doi: 10.1038/nm1591. Epub 2007 Jun 24. PMID 17589522
- [Background] Stahl A, Sapieha P, Connor KM, Sangiovanni JP, Chen J, Aderman CM, Willett KL, Krah NM, Dennison RJ, Seaward MR, Guerin KI, Hua J, Smith LE. Short communication: PPAR gamma mediates a direct antiangiogenic effect of omega 3-PUFAs in proliferative retinopathy. Circ Res. 2010 Aug 20;107(4):495-500. doi: 10.1161/CIRCRESAHA.110.221317. Epub 2010 Jul 15. PMID 20634487
- [Background] Smith LE. Through the eyes of a child: understanding retinopathy through ROP the Friedenwald lecture. Invest Ophthalmol Vis Sci. 2008 Dec;49(12):5177-82. doi: 10.1167/iovs.08-2584. Epub 2008 Aug 15. No abstract available. PMID 18708611
- [Background] SanGiovanni JP, Chew EY. The role of omega-3 long-chain polyunsaturated fatty acids in health and disease of the retina. Prog Retin Eye Res. 2005 Jan;24(1):87-138. doi: 10.1016/j.preteyeres.2004.06.002. PMID 15555528
- [Background] Pawlik D, Lauterbach R, Turyk E. Fish-oil fat emulsion supplementation may reduce the risk of severe retinopathy in VLBW infants. Pediatrics. 2011 Feb;127(2):223-8. doi: 10.1542/peds.2010-2427. Epub 2011 Jan 3. PMID 21199856
- [Background] Klein CJ, Havranek TG, Revenis ME, Hassanali Z, Scavo LM. Plasma fatty acids in premature infants with hyperbilirubinemia: before-and-after nutrition support with fish oil emulsion. Nutr Clin Pract. 2013 Feb;28(1):87-94. doi: 10.1177/0884533612469989. PMID 23319354
- [Background] Heird WC. The role of polyunsaturated fatty acids in term and preterm infants and breastfeeding mothers. Pediatr Clin North Am. 2001 Feb;48(1):173-88. doi: 10.1016/s0031-3955(05)70292-3. PMID 11236724
- [Background] O'Connor DL, Hall R, Adamkin D, Auestad N, Castillo M, Connor WE, Connor SL, Fitzgerald K, Groh-Wargo S, Hartmann EE, Jacobs J, Janowsky J, Lucas A, Margeson D, Mena P, Neuringer M, Nesin M, Singer L, Stephenson T, Szabo J, Zemon V; Ross Preterm Lipid Study. Growth and development in preterm infants fed long-chain polyunsaturated fatty acids: a prospective, randomized controlled trial. Pediatrics. 2001 Aug;108(2):359-71. doi: 10.1542/peds.108.2.359. PMID 11483801
- [Background] Fleith M, Clandinin MT. Dietary PUFA for preterm and term infants: review of clinical studies. Crit Rev Food Sci Nutr. 2005;45(3):205-29. doi: 10.1080/10408690590956378. PMID 16048149
- [Background] Smithers LG, Gibson RA, McPhee A, Makrides M. Effect of long-chain polyunsaturated fatty acid supplementation of preterm infants on disease risk and neurodevelopment: a systematic review of randomized controlled trials. Am J Clin Nutr. 2008 Apr;87(4):912-20. doi: 10.1093/ajcn/87.4.912. PMID 18400714
- [Background] Fewtrell MS, Morley R, Abbott RA, Singhal A, Isaacs EB, Stephenson T, MacFadyen U, Lucas A. Double-blind, randomized trial of long-chain polyunsaturated fatty acid supplementation in formula fed to preterm infants. Pediatrics. 2002 Jul;110(1 Pt 1):73-82. doi: 10.1542/peds.110.1.73. PMID 12093949
- [Background] Clandinin MT, Van Aerde JE, Merkel KL, Harris CL, Springer MA, Hansen JW, Diersen-Schade DA. Growth and development of preterm infants fed infant formulas containing docosahexaenoic acid and arachidonic acid. J Pediatr. 2005 Apr;146(4):461-8. doi: 10.1016/j.jpeds.2004.11.030. PMID 15812447
- [Background] Schulzke SM, Patole SK, Simmer K. Long-chain polyunsaturated fatty acid supplementation in preterm infants. Cochrane Database Syst Rev. 2011 Feb 16;(2):CD000375. doi: 10.1002/14651858.CD000375.pub4. PMID 21328248
- [Background] Born Too Soon | March of Dimes. March Dimes Found. Partnersh. Matern. Newborn Child Heal. Save Child. World Heal. Organ. 2012. Available at: http://www.marchofdimes.com/mission/global-preterm.aspx.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from October 2015 to November 2019 at University of California San Diego. Expectant parents of preterm infants were recruited and consented to the trial after admission to the hospital, either prior to or shortly after delivery.
Pre-assignment Details: 7 participants were consented but not assigned to an arm or group due to meeting exclusion criteria after birth -- 6 were consented before birth but were born over 30 weeks gestation, 1 had high liver function tests (LFTs) that were potentially indicative of liver disease.
Period: Overall Study
Arm/Group | Standard of Care (Standard Nutrition) | Omegaven
Started | 20 | 21
Completed | 17 | 10
Not Completed | 3 | 11
Not completed — Physician Decision | 1 | 7
Not completed — Hospital transfer | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (Standard Nutrition) | Omegaven | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Customized [Mean (Standard Deviation); unit: Gestational age (weeks)]
  Gestational age | 27.7 (1.7) | 27.2 (1.6) | 27.5 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 16 | 23
  Male | 13 | 5 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 12 | 21
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 6 | 11 | 17
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 5 | 6 | 11
Birth length [Mean (Standard Deviation); unit: centimeters] | 34.8 (3.4) | 33.7 (3.8) | 34.3 (3.6)
Birth head circumference [Mean (Standard Deviation); unit: centimeters] | 24.8 (2.0) | 24.8 (3.0) | 24.8 (2.5)
Birth weight [Mean (Standard Deviation); unit: grams] | 935 (239) | 914 (259) | 925 (246)

OUTCOME MEASURES:

1. Primary Outcome: Changes in mRNA Expression in Blood of STAT3, PPAR-ɣ, and STC-1 at T0
Description: Calculated using RNA extraction from blood, then quantitative polymerase chain reaction (qPCR) analysis.
  Biomarker significance:
  STAT3: role in hypoxia pathway leading to ROP (retinopathy of prematurity). Higher STAT3=greater ROP risk
  PPAR-ɣ: protective anti-angiogenic factor. Higher PPAR-ɣ=lower ROP risk
  STC-1: stress response protein. Higher STC-1=lower ROP risk
  Delta Ct meaning:
  qPCR gene expression analysis outputs Ct values for each genetic sample tested. A Ct value is the number of qPCR amplification cycles required for fluorescence, a proxy of gene expression, to cross a threshold. Lower Ct means less cycles of gene amplification needed for detectable fluorescence, therefore higher gene expression. Then target gene expression is calculated relative to a "housekeeping" control gene. Delta Ct=Ct(target gene)-Ct(control). Therefore, a HIGHER delta Ct value corresponds to a LOWER gene expression of the gene of interest relative to control.
Time Frame: T0 as defined in study protocol: prior to parental nutrition, within first three days of life
Population: Due to low RNA yield, we were unable to analyze all biomarkers of interest and could only analyze up to 3 biomarkers per sample. We chose to analyze STC-1 in the remaining batch of samples post-COVID-19 pandemic after updated literature review. This low RNA yield is why some groups below (e.g. Omegaven STC-1) have fewer analyzed blood samples than the other groups.
  One blood sample was analyzed per participant.
Measure: Mean (Standard Deviation); unit: delta Ct (amplification cycles)
Arm/Group | Standard of Care (Standard Nutrition) | Omegaven
Number analyzed (Participants) | 2 | 4
delta Ct (amplification cycles)
  STAT3 | 4.19 (1.72) | 7.58 (2.98)
  PPAR-gamma | 6.43 (2.17) | 11.32 (3.53)
  STC-1: number analyzed (Participants) | 2 | 3
  STC-1 | 22.21 (5.22) | 21.03 (3.90)
Statistical Analysis 1: Comparison: Standard of Care (Standard Nutrition) vs Omegaven; Null hypothesis: there was no difference in the average dCt values for relative gene expression of STAT-3 in T0 blood samples in the Standard of Care versus Omegaven group; Test type: Other — T-test for equality in means. The p-value threshold for significance was p < 0.05; p = 0.22, t-test, 2 sided
Statistical Analysis 2: Comparison: Standard of Care (Standard Nutrition) vs Omegaven; Null hypothesis: there was no difference in the average dCt values for relative gene expression of PPAR-gamma in T0 blood samples in the Standard of Care versus Omegaven group; Test type: Other — T-test for equality of means. The p-value threshold for significance was p < 0.05; p = 0.15, t-test, 2 sided
Statistical Analysis 3: Comparison: Standard of Care (Standard Nutrition) vs Omegaven; Null hypothesis: there was no difference in the average dCt values for relative gene expression of STC-1 in T0 blood samples in the Standard of Care versus Omegaven group; Test type: Other — T-test for equality of means. The p-value threshold for significance was p < 0.05; p = 0.78, t-test, 2 sided

2. Secondary Outcome: Pilot Assay of Basic Fatty Acid Concentrations in Blood at Time T2
Description: We measured concentrations of basic fatty acids in the blood plasma samples: eicosapentaenoic acid (EPA), docosahexaenoic acid (DHA), and arachidonic acid (AA). Blood samples were processed by the University of California San Diego lipidomics core and fatty acid concentrations in pmol/ml plasma were determined using gas chromatography-mass spectrometry.
Time Frame: T2 as defined in study protocol: 5 days after enteral nutrition full feeds have arrived; grace period +/-3 days therefore total 2-8 days after full enteral nutrition arrived.
Population: As stated in limitations or caveats, due to delays caused by the COVID-19 pandemic, funding limitations, and a clinical assessment of ROP outcomes in standard of care versus Omegaven infants, we elected to not conduct full fatty acid analyses for our remaining samples. As a result this data is only a pilot analysis and participant numbers were limited, and we could not conduct reliable statistical analyses for this outcome.
Measure: Mean (Standard Deviation); unit: pmol/ml plasma
Arm/Group | Standard of Care (Standard Nutrition) | Omegaven
Number analyzed (Participants) | 1 | 4
pmol/ml plasma
  EPA | 6826 (NA) — 1 participant (see analysis population description) | 132669 (19088)
  DHA | 61541 (NA) — 1 participant (see analysis population description) | 229583 (32725)
  AA | 334721 (NA) — 1 participant (see analysis population description) | 345122 (67435)

3. Secondary Outcome: Percentage of Eyes at the Furthest Stage of ROP Achieved
Description: Furthest severity stage of ROP achieved by patients in Arm 1 compared to Arm 2, per eye as assessed by weekly ROP screenings from approximately 31 weeks through 40 weeks adjusted age.
  Severity staging was determined in an eye exam per accepted clinical guidelines by a trained clinician and retinopathy of prematurity specialist. Briefly, staging is assigned based on the junction of the vascularized and avascular retina when viewed using indirect ophthalmoscopy. The higher the stage, the more severe the ROP. Per the American Association for Pediatric Ophthalmology and Strabismus,
  * Stage 0: no clear demarcation line between vascularized and non-vascularized retina
  * Stage 1: demarcation line that separates normal from premature retina
  * Stage 2: ridge with height and width
  * Stage 3: growth of fragile new abnormal blood vessels
Time Frame: approximately 31 to 40 weeks (adjusted age = gestation + post-natal age)
Population: As noted previously, 21 patients were enrolled in the Omegaven group, however for outcomes only 20 were analyzed because 1 patient was dropped from the study immediately after enrollment (deemed by the physician to be too sick from anemia and never started Omegaven).
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Standard of Care (Standard Nutrition) | Omegaven
Number analyzed (Participants) | 20 | 20
Number analyzed (eyes) | 40 | 40
percentage of eyes
  Stage 0 | 76.3 | 42.1
  Stage 1 | 5.3 | 7.9
  Stage 2 | 18.4 | 26.3
  Stage 3 | 0 | 23.7

4. Secondary Outcome: Number of Patients Requiring Laser Treatment in Arm 1 Versus Arm 2
Description: Number of patients with retinopathy of prematurity severe enough to require laser treatment by the adjusted age of 40 weeks, as assessed by weekly ROP screenings from approximately 31 weeks through 40 weeks adjusted age.
Time Frame: approximately 31 to 40 weeks (adjusted age = gestation + post-natal age)
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (Standard Nutrition) | Omegaven
Number analyzed (Participants) | 20 | 20
Participants | 0 | 5

5. Primary Outcome: Changes in mRNA Expression in Blood of STAT3, PPAR-ɣ, and STC-1 at T1
Description: as for outcome 1
Time Frame: T1 as defined in study protocol: 5 days after parenteral nutrition is started; grace period +/-3 days therefore total 2-8 days after parenteral nutrition started.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: delta Ct (amplification cycles)
Arm/Group | Standard of Care (Standard Nutrition) | Omegaven
Number analyzed (Participants) | 7 | 7
delta Ct (amplification cycles)
  STAT3 | 5.28 (4.79) | 6.98 (1.95)
  PPAR-gamma | 8.60 (5.38) | 10.51 (3.44)
  STC-1: number analyzed (Participants) | 5 | 6
  STC-1 | 20.73 (6.98) | 23.09 (4.02)
Statistical Analysis 1: Comparison: Standard of Care (Standard Nutrition) vs Omegaven; Null hypothesis: there was no difference in the average dCt values for relative gene expression of STAT-3 in T1 blood samples in the Standard of Care versus Omegaven group; Test type: Other — T-test for equality of means. The p-value threshold for significance was p < 0.05; p = 0.43, t-test, 2 sided
Statistical Analysis 2: Comparison: Standard of Care (Standard Nutrition) vs Omegaven; Null hypothesis: there was no difference in the average dCt values for relative gene expression of PPAR-gamma in T1 blood samples in the Standard of Care versus Omegaven group; Test type: Other — T-test for equality of means. The p-value threshold for significance was p < 0.05; p = 0.44, t-test, 2 sided
Statistical Analysis 3: Comparison: Standard of Care (Standard Nutrition) vs Omegaven; Null hypothesis: there was no difference in the average dCt values for relative gene expression of STC-1 in T1 blood samples in the Standard of Care versus Omegaven group; Test type: Other — T-test for equality of means. The p-value threshold for significance was p < 0.05; p = 0.50, t-test, 2 sided

6. Primary Outcome: Changes in mRNA Expression in Blood of STAT3, PPAR-gamma, and STC-1 at T2
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: delta Ct (amplification cycles)
Arm/Group | Standard of Care (Standard Nutrition) | Omegaven
Number analyzed (Participants) | 3 | 7
delta Ct (amplification cycles)
  STAT3 | 11.12 (2.80) | 4.66 (1.51)
  PPAR-gamma | 18.67 (3.64) | 7.31 (3.55)
  STC-1: number analyzed (Participants) | 2 | 6
  STC-1 | 28.42 (3.10) | 18.66 (3.87)
Statistical Analysis 1: Comparison: Standard of Care (Standard Nutrition) vs Omegaven; Null hypothesis: there was no difference in the average dCt values for relative gene expression of STAT-3 in T2 blood samples in the Standard of Care versus Omegaven group; Test type: Other — T-test for equality of means. The p-value threshold for significance was p < 0.05; p = 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Standard of Care (Standard Nutrition) vs Omegaven; Null hypothesis: there was no difference in the average dCt values for relative gene expression of PPAR-gamma in T2 blood samples in the Standard of Care versus Omegaven group; Test type: Other — T-test for equality of means. The p-value threshold for significance was p < 0.05; p = 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Standard of Care (Standard Nutrition) vs Omegaven; Null hypothesis: there was no difference in the average dCt values for relative gene expression of STC-1 in T2 blood samples in the Standard of Care versus Omegaven group; Test type: Other — T-test for equality of means. The p-value threshold for significance was p < 0.05; p = 0.01, t-test, 2 sided

7. Primary Outcome: Changes in mRNA Expression in Blood of STAT3 and PPAR-ɣ at T3
Description: Calculated using RNA extraction from blood, then quantitative polymerase chain reaction (qPCR) analysis.
  Biomarker significance:
  STAT3: role in hypoxia pathway leading to ROP (retinopathy of prematurity). Higher STAT3=greater ROP risk
  PPAR-ɣ: protective anti-angiogenic factor. Higher PPAR-ɣ=lower ROP risk
  Delta Ct meaning:
  qPCR gene expression analysis outputs Ct values for each genetic sample tested. A Ct value is the number of qPCR amplification cycles required for fluorescence, a proxy of gene expression, to cross a threshold. Lower Ct means less cycles of gene amplification needed for detectable fluorescence, therefore higher gene expression. Then target gene expression is calculated relative to a "housekeeping" control gene. Delta Ct=Ct(target gene)-Ct(control). Therefore, a HIGHER delta Ct value corresponds to a LOWER gene expression of the gene of interest relative to control.
Time Frame: T3 as defined in study protocol: Prior to discharge from hospital coinciding with time that ROP may be present, ≥35 weeks adjusted age.
Population: Due to low RNA yield and significant participant drop-out by the final time point, we only had one participant from the Omegaven group with a T3 blood sample that yielded enough RNA for gene expression analyses. As a result we were limited to analyzing only PPAR-gamma and STAT-3 and were unable to conduct statistical analyses on this time point.
  One blood sample was analyzed per participant.
Measure: Mean (Standard Deviation); unit: delta Ct (amplification cycles)
Arm/Group | Standard of Care (Standard Nutrition) | Omegaven
Number analyzed (Participants) | 5 | 1
delta Ct (amplification cycles)
  STAT3 | 3.90 (1.71) | 9.94 (NA) — only 1 participant (see above)
  PPAR-gamma | 9.15 (3.16) | 16.11 (NA) — only 1 participant (see above)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected while patients were actively enrolled in the study from October 2015 to December 2019. Each participant was assessed for adverse events for the duration of their active participation in the study, from 0-7 days of life until 40 weeks adjusted age (or withdrawal if prior to study completion).
Arm/Group | Standard of Care (Standard Nutrition) | Omegaven
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 2/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (Standard Nutrition) (N=20) | Omegaven (N=21)
Omegaven infusion rate discrepancy (Surgical and medical procedures) | 0 (0) | 1 (1) — 11/6/2016: HAL (hyperalimentation and intralipids) and Omegaven drips were hung but infusion rates were interchanged. Both drips were stopped and IV fluids without lipids were hung per physician orders.
Necrotizing enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (2) — Infant had NEC for which exploratory laparotomy and ileostomy were created. Reported because infant was receiving omegaven as part of the study but is not outside the complications of premature birth.

LIMITATIONS AND CAVEATS:
Due to the pandemic, we experienced significant delays in sample analysis. Upon resuming, due to limited funding, we decided not to conduct lipid analyses in remaining samples. Subject withdrawals, slower than expected recruitment and financial plan for batch testing may have also contributed to sample degradation. With low RNA yield, only a small number of samples were available for gene expression analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT02486042/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT02486042/ICF_001.pdf